CLINICAL TRIAL: NCT03867617
Title: A Prospective Controlled Trial to Evaluate Safety and Efficacy of in Vitro Expanded Recipient Regulatory T Cell Therapy and Tocilizumab Together With Donor Bone Marrow Infusion in HLA-mismatched Living Donor Kidney Transplant Recipients
Brief Title: Cell Therapy for Immunomodulation in Kidney Transplantation
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Thomas Wekerle (Other)
Collaborators: University Hospital Regensburg (Other)
Responsible Party: Sponsor-Investigator, Thomas Wekerle, Professor of Transplantation Immunology, Medical University of Vienna
Organization: Medical University of Vienna (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Trex001
Record Dates: First submitted 2019-03-06; First posted 2019-03-08 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Kidney Transplantation
MeSH Terms: interventions — tocilizumab; Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Study group (Experimental): Treatment with regulatory T cells, donor bone marrow and tocilizumab in addition to immunosuppressive drug therapy in kidney transplant recipients
  Interventions: Other: Regulatory T cells; Drug: Tocilizumab; Other: Bone marrow; Procedure: Kidney transplant; Other: Immunosuppressive drug therapy
- Control group (Active Comparator): Immunosuppressive drug therapy without treatment with regulatory T cells, donor bone marrow and tocilizumab in kidney transplant recipients
  Interventions: Procedure: Kidney transplant; Other: Immunosuppressive drug therapy

INTERVENTIONS:
Other: Regulatory T cells — Single infusion of expanded regulatory T cells.
  Arms: Study group
Drug: Tocilizumab — Treatment during first month post-transplant.
  Arms: Study group
Other: Bone marrow — Infusion of donor bone marrow cells.
  Arms: Study group
Procedure: Kidney transplant — Living donor kidney transplantation.
Other: Immunosuppressive drug therapy — Immunosuppressive drug therapy.

SUMMARY:
This study investigates treatment with recipient regulatory T cells and donor bone marrow together with tocilizumab for immunomodulation in living donor kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* Patient has provided written informed consent.
* Patient is 18 years or older.
* Patient is a planned recipient of a living donor kidney transplant.
* Patient is a planned recipient of an ABO blood group-compatible kidney graft.
* Patient is a planned recipient of a kidney graft from a donor that is not HLA (human leukocyte antigen)-identical.
* Patient is negative for DSA (donor-specific antibodies).
* WOCBP (women of child-bearing potential) must have a negative pregnancy test at inclusion.
* WOCBP must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 12 weeks after the study in such a manner that the risk of pregnancy is minimized.

Exclusion Criteria:

* Patient is EBV (epstein barr virus)-negative on serology.
* Patient is HIV-positive or suffering from chronic viral hepatitis.
* Patient is CMV (cytomegalo virus)-negative and receiving a kidney from a CMV-positive donor.
* Positive T-cell lymphocytotoxic cross match.
* Patient with prior kidney transplant or non-renal solid organ transplant.
* Patient has a known contraindication to any of the protocol-specified treatments.
* Patient had been diagnosed with a malignancy within 5 years prior to study entry, excluding non-metastatic basal or squamous cell carcinoma of the skin.
* Female patients who are breast-feeding.
* Female patients with a positive pregnancy test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Safety measured as GVHD (graft-versus-host disease), impaired graft function or patient death | 12 months
  Incidence of composite safety endpoint by 12 months post-transplant.
Chimerism | 1 month
  Total leukocyte donor chimerism in blood.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Wekerle, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna/Vienna General Hospital, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Oberbauer R, Edinger M, Berlakovich G, Kalhs P, Worel N, Heinze G, Wolzt M, Lion T, Wekerle T. A Prospective Controlled Trial to Evaluate Safety and Efficacy of in vitro Expanded Recipient Regulatory T Cell Therapy and Tocilizumab Together With Donor Bone Marrow Infusion in HLA-Mismatched Living Donor Kidney Transplant Recipients (Trex001). Front Med (Lausanne). 2021 Jan 27;7:634260. doi: 10.3389/fmed.2020.634260. eCollection 2020. PMID 33585521